CLINICAL TRIAL: NCT03401528
Title: A Single-blind, Randomized, Placebo-controlled, Phase 1, Single Ascending-dose and Repeat-dose, Safety and Tolerability Study of Intravenous AVB-S6-500 in Healthy Subjects
Brief Title: A Phase 1 AVB-S6-500 Safety and Tolerability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aravive, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: AVB500-HV-001
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — AVB-500 fusion protein

STUDY DESIGN:
Intervention Model Description: This study has two portions: a single ascending dose (SAD) portion consisting of 4 sequential dose escalation cohorts, and a repeat dose (RD) portion. In both study portions, subjects are randomized to receive either a study intervention (AVB-S6-500) or a placebo.
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose - AVB-S6-500 (Experimental): Four sequential dose escalation cohorts - patients are randomized either to investigational drug or matching placebo
  Interventions: Drug: AVB-S6-500
- Single Ascending Dose - placebo (Placebo Comparator): Four sequential dose escalation cohorts - patients are randomized either to investigational drug or matching placebo
  Interventions: Other: Placebo
- Repeat Dose - AVB-S6-500 (Experimental): Four single doses of the investigational drug or matching placebo - patients are randomized either to investigational drug or matching placebo
  Interventions: Drug: AVB-S6-500
- Repeat Dose - placebo (Placebo Comparator): Four single doses of the investigational drug or matching placebo - patients are randomized either to investigational drug or matching placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AVB-S6-500 — AVB-S6-500 is an investigational drug.
  Other Names: AVB500
  Arms: Repeat Dose - AVB-S6-500; Single Ascending Dose - AVB-S6-500
Other: Placebo — Matching placebo
  Arms: Repeat Dose - placebo; Single Ascending Dose - placebo

SUMMARY:
This is a randomized single-blind, placebo-controlled, Phase 1, single ascending dose (SAD) and repeat dose (RD), safety and tolerability study of AVB-S6-500 in healthy subjects. A SAD portion of the study consists of 4 sequential dose escalation cohorts, whereas RD portion of the study consists of a single cohort receiving 4 weekly doses of AVB-S6-500. In both SAD and RD study arms, subjects are randomized to receive either a study intervention (AVB-S6-500) or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female
* Age 18 - 55
* Body mass index (BMI) ranging between 18 and 30 kg/m2, inclusive
* Negative urine drug screen/alcohol breathalyzer results at Screening and at Day -1
* Has not used tobacco products during the 3 months prior to Screening and agrees to refrain from use throughout the study duration
* Female subjects of child-bearing potential must agree to use one of the study-approved effective contraceptive methods for the duration of the study and through 1 month after completion of the final study visit
* Male subjects must be either surgically sterilized or agree to use study-approved effective contraceptive methods for the duration of the study and through 1 month after completion of the final study visit
* If female, a negative serum pregnancy test at Screening and urinary pregnancy test at Day -1 is required
* Able to read, understand, and provide signed informed consent
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion Criteria:

* Blood pressure ≥ 140/90 mmHg or pulse > 100 beats/minute at Screening
* QTc intervals corrected for heart rate via the Fridericia method (QTcF) > 450 msec (males) and > 480 msec (females) at Screening
* Pregnant or a nursing female
* Male with a pregnant partner
* Currently enrolled in another clinical trial or has received treatment with an investigational drug during the 30 days (or 5 half-lives, whichever is longer) prior to dosing
* History of substance or alcohol abuse or dependency within the past
* Used any medications or over the-counter products within 14 days or 5 half lives (whichever is longer) prior to administration of study medication, including analgesics, hormonal contraceptives (oral contraceptive pills or implant), natural food supplements, or dietary or herbal supplements including vitamins)
* Donated blood in excess of 500 mL within 56 days prior to the dosing or intention of donating during the study through the month after completing the study
* Positive test results for hepatitis B virus (HBV) surface antigen, hepatitis C virus antibody (HCV), or human immunodeficiency virus (HIV)
* History or presence of any condition that, in the opinion of the Investigator, could interfere with the study conduct or observation
* A medical history of or any current clinically significant disorder, including but not limited to: asthma, angioedema, bronchospasm, ulcer disease, gastrointestinal bleeding, coagulation defects, hypertension, edema, heart failure, hypokalemia, cardiovascular disease, hypersensitivity reaction to any biologic drug, significant dermatologic diseases or condition that would significantly influence the immune response
* A serious illness, medical surgical procedure, or trauma resulting in missed work or hospitalization within the 30 days preceding the beginning of study treatment
* Received treatment for any type of cancer within the 5 years prior to enrollment
* An employee, family member, or student of the Investigator or clinical site

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AVB-S6-500 - Adverse events | Up to 6 weeks
  Monitoring of adverse events
Safety and tolerability of AVB-S6-500 - ECG | Up to 6 weeks
  Monitoring of 12 lead ECGs
Safety and tolerability of AVB-S6-500 -physical examination | Up to 6 weeks
  Physical examination of body systems
Safety and tolerability of AVB-S6-500 - vital sign | Up to 6 weeks
  Vital sign measurment
Safety and tolerability of AVB-S6-500 - clinical laboratory assessments | Up to 6 weeks
  Routine lab hematology, serum chemistry and coagulation

SECONDARY OUTCOMES:
AUC | Up to 6 weeks
  Area under the curve
Cmax | Up to 6 weeks
  Maximum observed concentration
Ctrough | Up to 6 weeks
  Serum concentration observed at end of a single dose and observed pre-dose during repeat doses
Tmax | Up to 6 weeks
  Time to reach maximum observed plasma concentration
λz | Up to 6 weeks
  Terminal phase elimination rate constant
t1/2 | Up to 6 weeks
  Terminal half-life
CL | Up to 6 weeks
  The total body clearance
V | Up to 6 weeks
  Volume of distribution
Pharmacodynamic parameter | Up to 6 weeks
  Concentration of the drug target

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Marbury, MD, Principal Investigator — Orlando Clinical Research Center
Locations (1):
- Orlando Clinical Research Center, Orlando, Florida, United States